CLINICAL TRIAL: NCT03821714
Title: Effects of Glucocorticoid Combined With Vitamin C and Vitamin B1 Versus Hydrocortisone Alone on Microcirculation in Severe Septic Shock
Brief Title: Effects of Glucocorticoid Combined With Vitamin C and Vitamin B1 on Microcirculation in Severe Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018ZDSYLL057-Y01
Record Dates: First submitted 2019-01-19; First posted 2019-01-30 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Septic Shock
Keywords: septic shock; glucocorticoid; vitamin C; microcirculation; Vitamin B1
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone; Ascorbic Acid; Thiamine; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid combination therapy Group (Experimental): Hydrocortisone 200mg continuous intravenous infusion(24h) combined with vitamin C1.5g intravenous infusion every 6 hours and vitamin B1 200mg intravenous infusion every 12 hours.
  Interventions: Drug: Glucocorticoid combination therapy
- Glucocorticoid Group (Active Comparator): Hydrocortisone 200mg continuous intravenous infusion(24h)
  Interventions: Drug: Glucocorticoid

INTERVENTIONS:
Drug: Glucocorticoid combination therapy — Glucocorticoid combination therapy is defined as the combination of hydrocortisone, vitamin C, and vitamin B1.
  Other Names: Hydrocortisone, vitamin C and vitamin B1
  Arms: Glucocorticoid combination therapy Group
Drug: Glucocorticoid — The glucocorticoid group was defined as the use of hydrocortisone alone.
  Other Names: Hydrocortisone
  Arms: Glucocorticoid Group

SUMMARY:
This study aimed to investigate the effect of Glucocorticoid combined with vitamin C and vitamin B1 versus hydrocortisone alone on microcirculation in septic shock patients.

DETAILED DESCRIPTION:
This prospective, double-blind, randomized, controlled trial enrolled septic shock patients admitted to the intensive care unite of a tertiary teaching hospital. We randomly assigned the enrolled patients to the treatment group (hydrocortisone combined with vitamin C and vitamin B1 added to standard care) and the control group (hydrocortisone alone added to standard care) in a 1:1 ratio. The primary outcome was perfusion vascular density (PVD) at 24 hours after treatment. We used the sublingual microcirculation imaging system to monitor PVD. We further validated the primary outcome by observing differences in renal perfusion monitored by renal contrast-enhanced ultrasound (CEUS) between the treatment group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Septic shock
2. A dose of norepinephrine (>15ug/min)
3. Age ≥18 and ≤80 years old
4. Signing Informed Consent

Exclusion Criteria:

1. Meet the inclusion criteria for more than 12 hours
2. Clinician judges that corticosteroid therapy should not be used
3. Pregnant
4. Uncontrolled malignancy
5. Glucocorticoid therapy was used within seven days before admission.
6. Expected death within 24 hours
7. The sublingual microcirculation cannot be measured

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Perfused vessel density (PVD) | 24 hours after treatment
  Determinant of capillary diffusive capacity

SECONDARY OUTCOMES:
proportion of perfusion vessels | 24 hours after treatment
  sublingual microcirculation parameter
total vascular density | 24 hours after treatment
  sublingual microcirculation parameter
microvascular flow index | 24 hours after treatment
  sublingual microcirculation parameter
renal contrast-enhanced ultrasound parameters | 24 hours after treatment
  renal perfusion
lactate | 24 hours after treatment
  Tissue perfusion parameter

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, PhD, Principal Investigator — Southeast University
Locations (1):
- Nanjing Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No